CLINICAL TRIAL: NCT00632164
Title: Sympathetic and Parasympathetic Responses to Specific Chiropractic Adjustments of Subluxation of the Cervical and Thoracic Spine
Brief Title: Sympathetic and Parasympathetic Responses to Specific Chiropractic Adjustments
Status: Completed | Type: Observational
Sponsor: Sherman College of Straight Chiropractic (Other)
Responsible Party: Dr. Arlene Welch, SHerman College
Other Study IDs: 1-Welch
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2008-03-10 (Estimated); Status verified 2008-02

CONDITIONS: Autonomic Nervous System

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Cervical adjustments
- 2: Thoracic adjustments

SUMMARY:
A study to determine if a chiropractic adjustment in the cervical spine will effect the parasympathetics and a chiropractic adjustment in the thoracic spine will effect the sympathetics.

ELIGIBILITY:
Inclusion Criteria:

* age 25-55, asymptomatic

Exclusion Criteria:

* HBP, heart condition

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Random ages 25-55 asymptomatic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2005-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Blood Pressure, Pulse Rate, Heart Rate Variability

CONTACTS AND LOCATIONS:
Overall Officials: Arlene R Welch, BS, DC, Principal Investigator — Sherman College
Locations (1):
- Sherman College, Spartanburg, South Carolina, United States